Title: Study 1 Replication and Extension of Prior Work

NCT Number: NCT04166591

Document date: 12/24/2024

The objective of this study was to see whether autistic and non-autistic children learn new words when they are presented in one of two conditions: as part of speech directly addressed to the child (Addressed condition), as part of speech they overhear (Overheard condition). Children participated in the experimental task in both conditions (within-subject design). The method was a behavioral experiment in which children were exposed to a novel word (e.g., "toma") in the context of one of three objects. The exposure either occurred with the experimenter looking directly at the child (Addressed condition) or looking at another adult (Overheard condition). They were then shown the three objects and given a prompt to identify which object is labeled by the novel word (e.g., "where is the toma?"). Children's eye gaze was coded as a measure of which object they preferred to look at after the prompt. After a delay of a few minutes, the test was repeated as a measure of retention.

The primary dependent variable reported here is the number of children who look at the target object more than would be expected by chance for each of the first test and the retention test; because there are three objects, chance is 33.33%.

The primary statistical analysis involves asking whether children in each condition (Addressed or Overheard) look at the target significantly more than chance levels. Binomial tests are used to see if the number of children who do so is significantly greater than would be expected by chance.